CLINICAL TRIAL: NCT03756636
Title: "Underwater" Technique With Submucosal Solution of Viscose Solution -SIC 8000 (EleviewTM) - For Endoscopic Resection of Cole-rectal Polyps With Signs of Fibrosis. Pilot Study
Brief Title: "Underwater" Technique With Submucosal Solution of Viscose Solution -SIC 8000 (EleviewTM) - For Endoscopic Resection of Cole-rectal Polyps With Signs of Fibrosis.
Acronym: UEMREleview
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2046
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-09

CONDITIONS: Colo-rectal Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Underwater" mucosectomy (Other): "Underwater" mucosectomy with submucosal injection of viscous solution -SIC 8000 (EleviewTM)
  Interventions: Procedure: "Underwater" mucosectomy with submucosal injection of viscous solution -SIC 8000 (EleviewTM)

INTERVENTIONS:
Procedure: "Underwater" mucosectomy with submucosal injection of viscous solution -SIC 8000 (EleviewTM) — "Underwater" mucosectomy with submucosal injection of viscous solution -SIC 8000 (EleviewTM)

SUMMARY:
All procedures are performed in the investigator's outpatient gastroenterology and digestive endoscopy unit by experienced endoscopists in conventional mucosectomies of the lower intestinal tract.

Before the procedure each patient, a normal endoscopic procedure. At the site of the lesion the lumen will be completely decompressed with aspiration of the gas, and then again relaxed with the instillation of only water. The EleviewTM will be injected into the submucosa in such quantities as to obtain a satisfactory lift of the lesion. The lesion will then be removed with a diathermic loop, preferably en-bloc, and in any case up to macroscopic evidence of complete resection. All the removed material will be stored and sent to histological analysis. Tolerability score will be recorded during the procedure.

Any "bleeding" (both intra- and post-procedural), perforation, post-polypectomy syndrome, stenosis or death in the 6 months following the procedure will be born "complication".

A surveillance colonoscopy including biopsy sampling of the research site scheduled 6 months after the procedure

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years.
* Signing of informed consent.
* Possibility of being subjected to the diagnostic and therapeutic procedures of the study.
* Presence of colo-rectal polypoid lesions ≥ 15mm presenting macroscopic aspects of fibrosis as a consequence of previous incomplete treatments or biopsies or relapses after previous removal.

Exclusion Criteria:

* Highly indicative morphological characteristics of carcinoma with submucosal invasion (Ulceration, Pit Pattern Vn according to Kudo et al.18)
* Pregnancy or breastfeeding
* ASA> 3
* Unstable personality or unable to adhere to the protocol procedures.
* Inability to provide informed consent.
* Injury not reachable endoscopically.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Macroscopically complete resection rate | 6 Months
6-month recurrence rate; | 6 Months
Rate of adverse events (according to the lexiconA ASGE). | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Gastroenterology Department, Humanitas Research Hospital, Rozzano, Milano, Italy